CLINICAL TRIAL: NCT03049462
Title: The Physiological Responses and Adaptation of Brown Adipose Tissue to Chronic Treatment With Beta3-Adrenergic Receptor Agonists
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 170054; 17-DK-0054
Record Dates: First submitted 2017-02-09; First posted 2017-02-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Brown Adipose Tissue; Energy Expenditure; Energy Metabolism; Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — mirabegron; Hydroquinones; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Females taking 100 mg of mirabegron
  Interventions: Drug: Mirabegron
- Cohort 2A (Active Comparator): Males taking 200 mg mirabegron
  Interventions: Drug: Mirabegron
- Cohort 2B (Placebo Comparator): Males taking placebo drug
  Interventions: Other: B Complex Plus Vitamin C Tablets
- Cohort 3A (Active Comparator): Females taking 100 mg of mirabegron
  Interventions: Drug: Mirabegron
- Cohort 3B (Placebo Comparator): Females taking placebo drug
  Interventions: Other: B Complex Plus Vitamin C Tablets

INTERVENTIONS:
Drug: Mirabegron — Women will take 100mg daily for 4 weeks. Men will take 200mg daily for 4 weeks. The medication is available in 50 mg tablets.
  Arms: Cohort 1; Cohort 2A; Cohort 3A
Other: B Complex Plus Vitamin C Tablets — Males will be randomized to take placebo versus active drug (mirabegron). Those taking placebo will take 4 tablets each day to mirror to active group (taking 4 tablets of 50 mg each).
  Arms: Cohort 2B; Cohort 3B

SUMMARY:
Background:

Brown adipose tissue (BAT) is a type of fat in the body. It may prevent weight gain, improve insulin sensitivity, and reduce fatty liver. Researchers want to see if BAT helps the body burn energy.

Objective:

To learn more about how BAT works to burn energy.

Eligibility:

People ages 18-40 with a body mass index between 18 and 40

Design:

Participants will be screened with:

Medical history

Physical exam

Blood, urine, and heart tests

Dietitian interview

Participants will have an overnight baseline visit. This includes:

Repeats of screening tests

Exercise test

Scans. For one scan, a radioactive substance is injected into the arm.

FSIVGIT: An IV is inserted into veins in the right and left arms. Glucose and insulin are injected in one arm. Blood glucose and insulin levels are measured from the other.

Metabolic suite: Participants stay 18 19 hours in a room that measures their metabolic rate. Monitors on the body measure heart rate, movement, and temperature.

Optional fat biopsy: A small piece of tissue is removed with a needle.

Participants will take 2-4 pills daily for 4 weeks. All women will take the drug mirabegron. Men will be randomly get either the drug or a placebo.

All participants will have a visit after 2 weeks of the pills. They will repeat the screening tests.

Participants will have an overnight visit 2 weeks later. They will repeat the baseline tests.

Participants will keep food and medication diaries.

Participants will have a follow-up visit 2 weeks after stopping the pills. This includes heart tests.

DETAILED DESCRIPTION:
Study Description:

This study is intended to address questions about human brown adipose tissue (BAT). Specifically, we plan to visualize BAT activity with acute cold exposure during drug naive and drug experienced visits. Thus, we will be studying changes in BAT activity from a chronic dosage of mirabegron.

Objectives:

Cohort 1: To measure changes in BAT metabolic activity in women seen after four weeks of daily treatment with the beta3-AR agonist mirabegron.

Cohort 2: To measure changes in BAT metabolic activity in men seen after four weeks of daily treatment with 200 mg of the beta3-AR agonist mirabegron compared to placebo

Cohort 3: To compare the changes in insulin sensitivity in each woman after four weeks of daily treatment with 100 mg of the beta3-AR agonist mirabegron with the changes in insulin sensitivity in each woman after four weeks of daily treatment with placebo

Primary Endpoints:

Cohort 1: The change in detectable cold exposure induced BAT metabolic activity in women, as visualized by F-FDG PET/CT.

Cohort 2: The change in detectable cold exposure induced BAT metabolic activity, as visualized by 18F-FDG PET/CT

Cohort 3: The change in glucose infusion rate, as measured by the hyperinsulinemic euglycemic clamp, in women after four weeks of daily treatment with 100 mg of the beta3-AR agonist mirabegron with the change in glucose infusion rate after four weeks of daily treatment with placebo

Secondary Endpoints:

1. To identify changes in metabolic health arising from BAT activation and/or prolonged treatment with regular 100 mg (females) or 200mg (men) doses of mirabegron.
2. To determine if there is an interaction between (a) BMI and (b) age with respect to the capacity to increase BAT metabolic activity.
3. To describe the structural and physiological changes in the adipose tissue depots, including cell lineage, size, and inflammation.
4. To assess whether there are improvements in the liver, including reduced stiffness and quantity of hepatic fat.

ELIGIBILITY:
* INCLUSION CRITERIA

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

Cohort 1: (complete)

1. Female
2. Age 18-40 years
3. BMI 18.00-40.0 kg/m^2
4. Able to understand the research and willing to sign a written informed consent document

Cohort 2: (complete)

1. Male
2. Age 18-40 years
3. BMI 18.00-40.0 kg/m^2
4. Able to understand the research and willing to sign a written informed consent document

Cohort 3:

1. Female
2. Age 18-40 years
3. BMI 25.0-50.0 kg/m^2 or BMI > 18.5 kg/m^2 with PCOS diagnosis
4. Diagnosis of PCOS based on NIH Criteria; defined by the presence of both clinical and/or biochemical signs of hyperandrogenism and oligo- or chronic anovulation.
5. Women of childbearing potential must agree to use a highly effective method of birth control, confirmed by the Investigator, for at least 3 months prior to the first study visit and continuing throughout the study duration.

   a. Highly effective methods of birth control include:

   i. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal

   ii. Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, or implantable

   iii. Intrauterine device

   iv. Intrauterine hormone-releasing system

   v. Bilateral tubal occlusion

   vi. Sexual abstinence, i.e., refraining from heterosexual intercourse (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant)

   vii. Vasectomized sexual partner (provided that partner is the sole sexual partner of the study participant and that the vasectomized partner has received medical assessment of the surgical success)

   b. Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrhoeic for >=12 months prior to the planned date of enrollment without an alternative medical cause.
6. Insulin resistance defined by either

   1. HOMA-IR score > 5.9 OR
   2. HOMA-IR score > 2.8 and <5.9, with HDL <51 mg/dL OR
   3. Fasting Insulin > 10.6 microU/mL
7. Able to understand the research and willing to sign a written informed consent document

EXCLUSION CRITERIA

1. Hypersensitivity and associated allergic reactions to mirabegron (or similar drug substances or components)
2. Abnormal bladder function, diagnosis of bladder outlet obstruction, urinary incontinence, urgency, and urinary frequency or use of antimuscarinic medication to treat overactive bladder (OAB)
3. Type 1 or Type 2 Diabetes mellitus, fasting serum glucose >125 mg/dL, and/or an HbA1c test >6.5%
4. Hypertension, defined as blood pressure (Bullet)140/90 mmHg, based on WHO guidelines (https://www.who.int/news-room/fact-sheets/detail/hypertension)
5. Hypo- or hyper-thyroid disease (TSH >5.0, <0.4 miU/L) that is controlled for less than one year
6. Anemia, defined by hemoglobin < 11.3 g/dL (females) or < 13.8 g/dL (males); sickle cell anemia or other blood disorders; and/or wound healing problems
7. Cardiovascular disease, cardiac arrhythmias, orthostasis, unstable vasomotor system, or renal impairment
8. A clinically significant abnormal ECG and/or QTc interval above normal
9. Elevated liver enzymes with probable or diagnosed liver disease (other than fatty liver disease)
10. Psychological conditions such as claustrophobia, untreated clinical depression or anxiety, untreated bipolar disorders, or forms of mental incapacity that would be incompatible with safe and successful participation in this study
11. Recent history in last 4 weeks of any local or systemic infectious disease with fever or requiring antibiotics
12. Self-reported intolerance of cold that would prevent the individual from spending several hours in a chilled room with a cooling vest
13. Current use of any drugs known to:

    * have major drug-drug interactions with mirabegron
    * Prolong QT interval
    * Alter glucose metabolism or cause insulin resistance (in last six months)
    * Treat diabetes mellitus
    * Treat hypertension
    * Be drugs of abuse
14. Self-reported weight loss or weight gain > 5% in the preceding 6 months.
15. Pregnancy, childbirth within the last year, or breastfeeding in the past 12 months
16. Individuals who spend >70% of daily hours outdoors since the exposure to varied environmental temperatures will potentially impact the ability to influence and measure BAT activity.
17. Addiction to alcohol or substances of abuse within the last 5 years
18. Self-reported current alcohol consumption of more than 2 servings of alcohol per day
19. Self-reported current use of nicotine and/or tobacco products
20. Has participated in a clinical trial with an investigational or marketed drug within 2 months
21. Have had previous radiation exposure (X-rays, PET scans, etc.) within the last year or anticipate radiation exposure in the upcoming year - clinical and/or research - that would exceed research limits
22. Donated blood within last 2 months
23. Unwilling or unable to eat metabolic meals, as determined by dietitian consult.
24. Any other circumstances or criteria that would preclude safe participation in the study in the clinical judgment of the investigator

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Cohorts 1 and 2: Change in BAT metabolic activity | 4 weeks
  Change in brown adipose tissue (BAT) metabolic activity as measured by 18FFDG PET/CT
Cohort 3: Change in insulin sensitivity | 4 weeks
  Change in glucose infusion rate, as measured by the hyperinsulinemic euglycemic clamp

SECONDARY OUTCOMES:
Identify changes in metabolic health arising from BAT activation and/or prolonged treatment with mirabegron | 4 weeks
  Change in metabolic health parameters including body weight, fat mass, glucose tolerance, changes in levels of hormones, and improved liver function
Cohort 3: Changes in BAT metabolic activity | 4 weeks
  Change in brown adipose tissue (BAT) metabolic activity as measured by 18FFDG PET/CT
Cohorts 1 and 2: Changes in insulin sensitivity | 4 weeks
  Changes in glucose infusion rate, as measured by the hyperinsulinemic euglycemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Cypess, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: >With whom - Researchers who provide a methodologically sound proposal@@@@@@>For what types of analysis - To achieve aims in the approved proposal@@@@@@>By what mechanism will data be made available? - Proposals should be directed to aaron.cypess@nih.gov. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] O'Mara AE, Johnson JW, Linderman JD, Brychta RJ, McGehee S, Fletcher LA, Fink YA, Kapuria D, Cassimatis TM, Kelsey N, Cero C, Sater ZA, Piccinini F, Baskin AS, Leitner BP, Cai H, Millo CM, Dieckmann W, Walter M, Javitt NB, Rotman Y, Walter PJ, Ader M, Bergman RN, Herscovitch P, Chen KY, Cypess AM. Chronic mirabegron treatment increases human brown fat, HDL cholesterol, and insulin sensitivity. J Clin Invest. 2020 May 1;130(5):2209-2219. doi: 10.1172/JCI131126. PMID 31961826
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-DK-0054.html